CLINICAL TRIAL: NCT05448170
Title: Linerixibat Compassionate Use for Cholestatic Pruritus in Adult Patients With Primary Biliary Cholangitis
Brief Title: Linerixibat Compassionate Use for Cholestatic Pruritus Adult Patients With Primary Biliary Cholangitis (PBC)
Status: Available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 217327
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pruritus
Keywords: Linerixibat; Individual Patient Compassionate Use; Primary Biliary Cholangitis; Ileal bile acid transporter (IBAT) inhibitor
MeSH Terms: conditions — Pruritus; Liver Cirrhosis, Biliary

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Linerixibat — open label investigational product

SUMMARY:
The goal of this compassionate use program is to provide a mechanism to supply linerixibat, on an individual named patient basis. This program is for treatment of individuals who have cholestatic pruritus associated with PBC who are deemed at high risk of a significant clinical event as a result of their pruritus and for whom all available pharmaceutical treatment options for cholestatic pruritus have been unsuccessful or are considered to not be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cholestatic pruritus associated to PBC identified by their healthcare provider as being at high risk of a significant clinical event as a result of their pruritus.
* Male and female >= 18 years of age.
* Participants for whom all available pharmaceutical treatments for cholestatic pruritus in PBC have been unsuccessful or are considered to not be appropriate.
* Contraceptive/Barrier Requirements (applicable for female participants only): A female participant is eligible if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  1. Is not a woman of childbearing potential (WOCBP) OR
  2. Is a WOCBP and using an acceptable contraceptive method during the treatment with linerixibat and for at least 4 weeks after the last dose of linerixibat.

Exclusion Criteria:

* Advanced chronic liver disease (e.g. cirrhosis Child-Pugh C) or presence of hepatic decompensation (e.g. variceal bleeding, encephalopathy).
* Use of obeticholic acid or other IBAT inhibitor.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline